CLINICAL TRIAL: NCT04904497
Title: Early Occupational Therapy in Mechanical Ventilated Patients With Covid-19: Multicentre Pilot Randomized Clinical Trial
Brief Title: Early Occupational Therapy in Mechanical Ventilated Patients With Covid-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Hospital Base Valdivia (Unknown); Hospital Santiago Oriente - Dr. Luis Tisné Brousse (Unknown)
Responsible Party: Principal Investigator, Eduardo Tobar, Associated professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Reh-Covid-19
Record Dates: First submitted 2021-04-30; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Critical Illness; Impairment, Cognitive; Impairment, Coordination
MeSH Terms: conditions — COVID-19; Critical Illness; Cognitive Dysfunction; Ataxia

STUDY DESIGN:
Intervention Model Description: A control group (standard ASDM measures) or an intervention group (early and intensive occupational therapy + ASDM) will be randomized. The intervention group will receive 20 occupational therapy sessions. The interventions will be organized on the basis of i) level of sedation, ii) presence or absence of delirium (according to CAM ICU +/- (Confusion Assessment Method Intensive Care Unit)), iii) movement with or without gravity (cut-off point 3 points in elbow flexion movement in Medical Research Council(MRC)). The areas of intervention implemented by occupational therapist will be: i) Polysensory stimulation, ii) Cognitive stimulation, iii) Basic activities of daily living, iv) Motor function stimulation, v) Education
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, researchers, recruiters, evaluators, control group team and data analyst will be masked. These teams will not have contact with the interventionists of the experimental group. Evaluators who have contact with the patients of both groups, they will be professionals from other medical units, who do not know the ICU team, and will only be able to maintain their dialog, according to the guideline of each evaluation.
  It is not possible to mask the treating occupational therapist and patient receiving OT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Occupational Therapy (Experimental): These sessions will be implemented by occupational therapists trained in ICU, who will conduct 20 sessions of 30 min, distributed depending on the level of sedation, i) SAS (Sedation-Agitation Scale) 1 patients have one session each 48 h, evaluating the change of sedation level each 24 h; ii) SAS 2 patients have one session each 24 h, iii) SAS 3-5 have two sessions every day. The sessions will begin once the patient needs mechanical ventilation for at least 12 h
  Interventions: Behavioral: Early Occupational Therapy
- Standard (No Intervention): The ASDM protocol will be implemented to mechanically ventilated patients in the ICU, following the aspects recommended by experts and the current evidence. For this, the team of medical, nurses, and physiotherapist will be trained to understand and facilitate the ASDM actions that each one must implement.
  Occupational Therapy interventions for control group will be allowed for this group only before 1 week after the first day on light sedation

INTERVENTIONS:
Behavioral: Early Occupational Therapy — Occupational therapists will implement the following activities:
  * Polysensory stimulation: external stimulation for increasing the level of alertness. It will be implemented with SAS 2 one session each 24 h.
  * Cognitive stimulation: bundle of exercises for activating mental functions, i.e: alertness, visual perception, memory, calculus, problem solving, praxis, language. Patients with SAS 3, 4 and 5. In SAS <2, 6> environmental orientation will be considered
  * Basic activities of daily living (BADLs): promotion of independence that initially practice hygiene, personal grooming. Patients with SAS 3, 4 and 5
  * Motor function Stimulation: exercises to keep the patient's upper extremities active and functional. Patients with SAS with 3,4 and 5. Patients with SAS 1 and 2 will use adaptations to prevent edema and bedsores on vulnerable body areas
  * Education: trained family members and health staff about the intervention process
  Arms: Early Occupational Therapy

SUMMARY:
This study evaluates the feasibility of an early occupational therapy (OT) protocol in critical adult patients requiring mechanical ventilation with Covid-19.

DETAILED DESCRIPTION:
A randomized clinical trial with an experimental-control will be implemented, considering the prospective multicenter group, with parallel groups, in a 1:1 ratio, in 3 Chilean hospitals.

A control group will has a standard analgesia, sedation, delirium and mobilization (ASDM) measures or an intervention group will have early OT plus ASDM.

The intervention group will receive 20 OT sessions, which considers a predefined protocol of actions according to the patient's condition

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years.
* Need for hospitalization in ICU.
* At least 12 h of invasive mechanical ventilation
* Informed consent signed by legal representative and / or patient.
* Positive covid-19 diagnosis

Exclusion Criteria:

* Known cognitive impairment before admission with short IQCODE (Informant Questionnaire on Cognitive Decline in the Elderly) Scores> 3.3 were excluded.
* Previous functional impairment, FAQ (Functional Activities Questionnaire) defined as > 6 points.
* Severe communication disorder and cultural limitation of language (language different from Spanish)
* Patient with limited therapeutic proportionality.
* Neurocritical patients (moderate-severe Traumatic Brain Injury / stroke of some kind / among others)
* Spinal injury or unstable fractures that limit mobilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional independence at hospital discharge | Day 28 (+/- 3 days) from beginning of mechanical ventilation
  The FIM (Functional independence measure) instrument will be applied by evaluator team. This scale shows that higher score is better, which will be compared between control and experimental group

SECONDARY OUTCOMES:
Delirium-free days | Defined as the number of days in the first 14 days with the CAM-ICU instrument negative and non-coma day.
  CAM-ICU (Confusion Assessment Method Intensive Care Unit) instrument will be applied once a day by evaluatorhigher score is better, which will be compared between control and experimental group
Coma-free days | Defined as the number of days in the first 14 days with the SAS.
  SAS (Sedation-Agitation Scale) instrument will be applied once a day by evaluator. If SAS 1-2: coma day
Delirium-coma free days | Defined as the number of days in the first 14 days with the SAS and CAM-ICU
  SAS and CAM-ICU instruments will be applied once a day by evaluator. Every day without coma or delirium its an delirium-coma free day
Functional independence at hospital discharge | Day 90 (+/- 7 days) from beginning of mechanical ventilation
  The FIM (Functional independence measure) instrument will be applied by evaluator team. This scale shows that higher score is better, which will be compared between control and experimental group
Cognitive status of patients | Day 28 (+/- 3 days) from beginning of mechanical ventilation and day 90 (+/- 7 days)after hospital discharge
  MoCA (Montreal Cognitive Assessment) instrument (cognitive status).This scale shows that higher score is better, which will be compared between control and experimental group
Motor status of patients | Day 28 (+/- 3 days) from beginning of mechanical ventilation
  Grip strength (motor status) with dynamometer will be applied by evaluator. This scale shows that higher score is better, which will be compared between control and experimental group
Quality of life of patients | Day 90 (+/- 7 days) from beginning of mechanical ventilation
  EQ-5D-5L (Euro Qol 5 dimensions 5 level) will be applied by evaluator. It will be considered a cut-off point in the Chilean population
Characterization of occupational therapy interventions | Days of patient hospitalization
  Number of sessions implemented, number of sessions suspended

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No